CLINICAL TRIAL: NCT02892968
Title: ED Ultrasonographic Regional Anesthesia to Prevent Incident Delirium in Hip Fracture Patients (EDU-RAPID) Multi-center Stepped Wedge Cluster Randomized Trial
Brief Title: ED Ultrasonographic Regional Anesthesia to Prevent Incident Delirium in Hip Fracture Patients
Acronym: EDU-RAPID
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 201503MOP
Record Dates: First submitted 2016-08-09; First posted 2016-09-08 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: Hip Fractures; Delirium
Keywords: Regional Anesthesia Ultrasound guided; Emergency Department; Knowledge to Practice Intervention
MeSH Terms: conditions — Hip Fractures; Delirium; Emergencies

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- U/S Guided Regional Anesthesia (Experimental): Fascia-Iliaca Block(FIB) Femoral Nerve Block(FNB)
  All participating emergency physicians (EPs) will be randomly assigned to the order they receive training in a stepped wedge design. Thus all EPs will begin the trial as "control physicians". EPs will then be trained to use two approaches to ultrasound (U/S) guided regional anesthesia, the fascia iliaca and femoral nerve blocks. Which block that will be used will be randomly determined at the individual patient level
  Interventions: Procedure: Fascia-Iliaca Block(FIB); Procedure: Femoral Nerve Block(FNB)
- Current Local Standard Analgesia (No Intervention): All participating emergency physicians (EPs) will be randomly assigned to the order they receive training in a stepped wedge design. Thus all EPs will begin the trial as "control physicians". Physicians who are in the control group will provide current local standard of analgesic care for hip fracture patients such as the use of IV opiods with supplemental acetaminophen and non-steroidal anti-inflammatory agents until they receive training.

INTERVENTIONS:
Procedure: Fascia-Iliaca Block(FIB) — The target of the FIB is the potential space between the fascia iliaca and the iliacus muscle, at least 4 cm lateral to the Femoral artery. This is neither a drug nor a device.
  Arms: U/S Guided Regional Anesthesia
Procedure: Femoral Nerve Block(FNB) — The target of the FNB technique is the intersection of the fascia iliaca and the femoral nerve. This is neither a drug nor a device.
  Arms: U/S Guided Regional Anesthesia

SUMMARY:
Hip fractures are common, costly and affect older people - Canadians spend 1 billion dollars to treat hip fractures each year. Unfortunately, as many as two-thirds of hip fracture cases suffer a complication known as delirium, or acute confusion. Patients with delirium may become frightened and agitated. This in turn leads to other serious problems. Having delirium doubles the chances of dying or can increase the need for admission into a nursing home. People with delirium spend an extra week in hospital on average.

Using ultrasound to locate and 'freeze' or block specific nerves can stop hip fracture pain almost immediately, and use of this technique is known to reduce delirium when administered by Anaesthetists to patients at the time of their hip operation. Unfortunately, patients with hip fractures commonly wait hours or even days in the Emergency Department (ED) prior to their operation. Currently, these patients are given narcotic pain killers like morphine to dull their pain, as most ED physicians have not been trained in using this 'freezing' technique and Anaesthetists are rarely able to leave the operating room to administer freezing to patient in the ED.

The EDU-RAPID study will test whether training ED physicians on how to use the nerve freezing technique will reduce the number of patients who develop delirium after a hip fracture. To study this, ED physicians will be trained at 6 hospitals in small groups every 6 weeks over 18 months. The study will look at how patients who are treated by ED physician who has been trained compare to patients treated by a ED physician who has not yet been trained. Also, the study will see if the training motivates ED physicians to use the block regularly.

If correct, this study could significantly improve the comfort, quality of life, and independence of patients who suffer a hip fracture. In addition, if the study shows a reduction in delirium rates, this could represent a significant cost reduction to the health care system.

ELIGIBILITY:
Inclusion Criteria:

* At the cluster level, ED physicians practicing at a participating site will be eligible.
* At the patient level, all hip fractures seen by a participating ED physician will be eligible

Exclusion Criteria:

* ED physicians who work casually (less than 0.25 Full Time Equivalent)
* ED Physicians who are routinely using U/S guided RA for hip fracture patients, or decline participation in the trial.
* Patients' age less than 65 years;
* Patients who are delirious on initial assessment by ED physician or severe dementia
* Patients with communication problems (critically ill, unconscious, language barrier despite use of secure telephone-based translation service)
* Patients with allergies to narcotics or local anesthetic; or anticoagulant use (e.g. warfarin, dabigatran, rivaroxaban).
* Patients with hip fractures not requiring surgery (e.g. greater trochanter avulsion) will also be excluded.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2016-09; Primary Completion 2020-09 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Overall rate of incident delirium | Time of injury to post-injury day 7
Time to onset of incident delirium | Time of injury to post-injury day 7

SECONDARY OUTCOMES:
The rate of regional anesthesia use by intervention physicians for hip fracture patients | Time of injury to operation to maximum of 7 days
Time to perform the block | Time block started to completion to maximum of 2 hours
Pain Severity on 0-10 Numeric Rating Scale as assessed by treating MD or Nurse after administration of regional anesthesia | 30 minutes and 60 minutes after administration of regional anesthesia
Numeric Rating Scale (1-5) Effectiveness of block (pain reduction measured)at 30 minutes | 30 minutes after administration of regional anesthesia
Supplementary narcotic analgesics used pre-operatively, measured in morphine equivalent units | Time of Injury to operation measured to a maximum of 7 days
Maximum severity of delirium using the validated Delirium Index (DI) | Time of injury to post-injury day 7
Cognitive Assessment Method (CAM) status (CAM + or CAM -) measurement at hospital discharge | Admission to Discharge to a maximum of 100 days
Complications from the regional anesthesia including hematoma and persistent nervous dysfunction | Time of injury to post-injury day 7
Adverse events, including in-hospital falls, cardiovascular events and deaths; Hospital length of stay | Time of injury to 1 year follow-up
Functional status measured using Older Americans' Resources and Services (OARS) Activities of Daily Living Questionnaire at 1 month and 1 year follow-up | 1 month and 1 year follow-up from Time of Injury
Proportion of patients who return to independent living at discharge | Admission to Discharge to a maximum of 1 year
Mortality within 1 year post-operatively | 1 year follow-up from time of injury

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybrook Health Sciences Center, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee JS, Chenkin J, Simard R, Bhandari T, Woo MY, Perry JJ, Eagles D, Wong C, McRae AD, Lang E, Newbigging J, Sivilotti MLA, Chernoff I, Borgundvaag B, McLeod SL, Melady D, Kiss A, Emond M. Ultrasound-Guided Regional Anesthesia by Emergency Physicians for Hip Fractures and Delirium: A Randomized Clinical Trial. JAMA Netw Open. 2025 Dec 1;8(12):e2549337. doi: 10.1001/jamanetworkopen.2025.49337. PMID 41396601
- [Derived] Lee JS, Bhandari T, Simard R, Emond M, Topping C, Woo M, Perry J, Eagles D, McRae AD, Lang E, Wong C, Sivilotti M, Newbigging J, Borgundvaag B, McLeod SL, Melady D, Chernoff L, Kiss A, Chenkin J. Point-of-care ultrasound-guided regional anaesthesia in older ED patients with hip fractures: a study to test the feasibility of a training programme and time needed to complete nerve blocks by ED physicians after training. BMJ Open. 2021 Jul 5;11(7):e047113. doi: 10.1136/bmjopen-2020-047113. PMID 34226222
- [Derived] Guay J, Kopp S. Peripheral nerve blocks for hip fractures in adults. Cochrane Database Syst Rev. 2020 Nov 25;11(11):CD001159. doi: 10.1002/14651858.CD001159.pub3. PMID 33238043